CLINICAL TRIAL: NCT04956627
Title: A Phase 1, Single-Center, Parallel-Group, Open-Label, Randomized, Drug-Drug Interaction Study to Assess the Effect of Itraconazole, Phenytoin, and Gemfibrozil on the Pharmacokinetics of a Single Oral Dose of BMS-986166 in Healthy Participants
Brief Title: A Study to Assess the Effect of Itraconazole, Phenytoin and Gemfibrozil on the Drug Levels of BMS-986166 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IM018-004
Record Dates: First submitted 2021-07-01; First posted 2021-07-09 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; BMS-986166
MeSH Terms: interventions — BMS-986166; Itraconazole; Phenytoin; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986166 (Experimental)
  Interventions: Drug: BMS-986166
- BMS-986166 + Itraconazole (Experimental)
  Interventions: Drug: BMS-986166; Drug: Itraconazole
- BMS-986166 + Phenytoin (Experimental)
  Interventions: Drug: BMS-986166; Drug: Extended Phenytoin Sodium
- BMS-986166 + Gemfibrozil (Experimental)
  Interventions: Drug: BMS-986166; Drug: Gemfibrozil

INTERVENTIONS:
Drug: BMS-986166 — Specified dose on specified days
Drug: Itraconazole — Specified dose on specified days
  Other Names: Sporanox
  Arms: BMS-986166 + Itraconazole
Drug: Extended Phenytoin Sodium — Specified dose on specified days
  Other Names: Dilantin
  Arms: BMS-986166 + Phenytoin
Drug: Gemfibrozil — Specified dose on specified days
  Other Names: Lopid
  Arms: BMS-986166 + Gemfibrozil

SUMMARY:
The purpose of this study is to evaluate the effect of itraconazole, phenytoin and gemfibrozil on the drug levels of BMS-986166 and its active metabolite BMT-121795. Participants will be randomly assigned to one of four groups and will remain in the study clinic for the duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 55 kg.
* Body mass index (BMI) of 19.0 to 32.0 kg/m², inclusive. BMI = weight (kg)/(height [m])².
* Healthy female subjects of non-childbearing potential, or male subjects, as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations.

Exclusion Criteria:

* Any significant acute or chronic medical illness or any other condition listed as a contraindication in the itraconazole, phenytoin, or gemfibrozil package inserts.
* History of any type of heart disease, including ischemia, infarction, clinically significant arrhythmias, sinus syndrome, hypertension, symptomatic orthostatic hypotension, atrioventricular block of any degree, bradycardia, syncope, clinically significant 12-lead ECG abnormalities, or any congenital heart disease.
* History of stroke or transient ischemic attacks.
* History of asthma or chronic obstructive pulmonary disease diagnosed or treated within the past 5 years.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986166 | Up to Day 22
Cmax of BMT-121795 | Up to Day 22
Time of maximum observed plasma concentration (Tmax) of BMS-986166 | Up to Day 22
Tmax of BMT-121795 | Up to Day 22
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of BMS-986166 | Up to Day 22
AUC(0-T) of BMT-121795 | Up to Day 22
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF))of BMS-986166 | Up to Day 22
AUC(INF) of BMT-121795 | Up to Day 22
Terminal plasma half-life (T-HALF) of BMS-986166 | Up to Day 22
T-HALF of BMT-121795 | Up to Day 22
Apparent total body clearance (CL/F) of BMS-986166 | Up to Day 22
Apparent volume of distribution (Vz/F) of BMS-986166 | Up to Day 22
Ratio of BMT-121795 Cmax to parent Cmax corrected for molecular weight (MR_Cmax) | Up to Day 22
Ratio of BMT-121795 AUC(0-T) to parent AUC(0-T) corrected for molecular weight (MR_AUC(0-T)) | Up to Day 22
Ratio of BMT-121795 AUC(INF) to parent AUC(INF) corrected for molecular weight (MR_AUC(INF)) | Up to Day 22

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 55
Number of participants with Serious Adverse Events (SAEs) | Up to Day 55
Number of participants with physical examination abnormalities | Up to Day 55
Number of participants with clinically significant changes in vital signs: Body temperature | Up to Day 55
Number of participants with clinically significant changes in vital signs: Respiratory rate | Up to Day 55
Number of participants with clinically significant changes in vital signs: Blood pressure | Up to Day 55
Number of participants with clinically significant changes in vital signs: Heart rate | Up to Day 55
Number of participants with clinically significant changes in ECG parameters: PR interval | Up to Day 55
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Number of participants with clinically significant changes in ECG parameters: QRS | Up to Day 55
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Number of participants with clinically significant changes in ECG parameters: QT interval | Up to Day 55
  The QT interval is the time from the start of the Q wave to the end of the T wave
Number of participants with clinically significant changes in ECG parameters: QTcF | Up to Day 55
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Number of participants with clinically significant changes in laboratory values: Hematology tests | Up to Day 55
Number of participants with clinically significant changes in laboratory values: Chemistry tests | Up to Day 55
Number of participants with clinically significant changes in laboratory values: Urinalysis | Up to Day 55

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Hassman Research Institute, Berlin, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm